CLINICAL TRIAL: NCT01372111
Title: Chemoradiotherapy With Very Low Dose Elective Nodal IMRT for Locally Advanced Head & Neck Cancer: the CCRO11 Multi-Institutional Phase II Trial
Brief Title: Chemoradiotherapy With Elective Low Dose Nodal Radiation for Locally Advanced Head and Neck Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Coastal Carolina Radiation Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); New Hanover Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCRO11; U54CA142152-02 (NIH)
Record Dates: First submitted 2011-06-06; First posted 2011-06-13 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Head and Neck Cancer
Keywords: Stg III or IVa Squamous Cell Carcinoma.; Advanced
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 35 mg/m2 IV weekly during weeks 1 through 6 of IMRT.
  Other Names: Cis-Diamminedichloroplatinum, DDP
Radiation: Elective Nodal Irradiation (ENI) — Low risk planning target volume (PTV) of 36 Gy at 2 Gy per fraction daily to bilateral, uninvolved neck nodal regions at risk for harboring microscopic cancer. High risk PTV will receive 70 Gy.

SUMMARY:
Concurrent chemotherapy and radiation therapy (chemoRT) has become the standard of care for treatment of many patients with advanced head and neck squamous cell carcinoma (HNSCC), though many clinical questions remain. Prior experience has revealed locoregional control (LRC), disease free survival (DFS) and overall survival (OS) at 3 years exceeding 80% after treatment with the use of hyperfractionated intensity modulated radiation therapy (IMRT) and concurrent weekly cisplatin chemotherapy for patients with locally advanced HNSCC. This multi-institutional phase II ZCC00204 trial resulted in an acceptable quality of life (QOL) and toxicity profile. The current trial is an attempt to maintain high LRC, while further minimizing both acute and chronic toxicities, and maximizing QOL.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven squamous cell carcinoma of oral cavity, oropharynx, hypopharynx, or larynx
* No surgical resection of primary site or neck dissection (excisional biopsy of lymph node is permitted)
* Human Papilloma Virus (HPV) testing of tumor performed; HPV p16 by immunohistochemistry
* Stage III or IVa disease (T1-2N1-3M0, T3-4N0-3M0) excluding T1-2N1 oral cavity and tonsil primaries and any N2C or bilateral N3 disease. Patients with T2N0 cancer of the base of tongue and hypopharynx are eligible
* ECOG performance status 0-1
* Age >18 years
* No current pregnancy
* No other invasive malignancies within the last 2 years Patients with basal cell or squamous cell skin cancers or carcinoma in situ of any site are eligible.
* No prior radiotherapy to the head and neck region
* No prior cisplatin chemotherapy
* No symptomatic coronary disease or myocardial infarction within the last 6 months
* Laboratory evaluation: ANC > 2,000/mm3, platelets >100,000/mm3, creatinine < 1.5 mg/dl, creatinine clearance > 50 ml/min, bilirubin < 1.5 mg/dl, AST or ALT < 2X upper normal limit
* Study-specific consent signed prior to entry

Exclusion Criteria:

* Second primary malignancy that is clinically detectable
* Inability or unwillingness to comply with chemoRT
* Prior radiotherapy, chemotherapy, or investigational treatment for squamous cell carcinoma of head and neck.
* Metastatic disease (M1)
* Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2011-03; Primary Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
To assess the actuarial elective nodal failure (ENF) rate for patients with locally advanced HNSCC treated with chemoRT including very low dose elective nodal IMRT and concurrent weekly cisplatin. | 4 years

SECONDARY OUTCOMES:
To assess actuarial LRC, DFS, and OS rates. | 4 years
To evaluate patients' quality of life (QOL). | 4 years
To evaluate grade 3-5 toxicity by CTCAE v4.0, with special attention to swallowing function, feeding tube dependence, and xerostomia. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Patrick D. Maguire, M.D., Principal Investigator — Coastal Carolina Radiation Oncology
Locations (5):
- United States (5):
  - Coleman Radiation Oncology Center, Morehead City, North Carolina
  - CarolinaEast Cancer Care, New Bern, North Carolina
  - South Atlantic Radiation Oncology, Supply, North Carolina
  - Coastal Carolina Radiation Oncology, Wilmington, North Carolina
  - Zimmer Cancer Center, Wilmington, North Carolina

REFERENCES:
- [Result] Maguire PD, Papagikos M, Hamann S, Neal C, Meyerson M, Hayes N, Ungaro P, Kotz K, Couch M, Pollock H, Tepper J. Phase II trial of hyperfractionated intensity-modulated radiation therapy and concurrent weekly cisplatin for Stage III and IVa head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2011 Mar 15;79(4):1081-8. doi: 10.1016/j.ijrobp.2009.12.046. Epub 2010 Apr 8. PMID 20378262